CLINICAL TRIAL: NCT06165068
Title: Effects of Antiplatelet and Antioxidant Agents on Drusen Progression: A Pilot, Prospective Cohort Study
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Navamindradhiraj University (Other)
Responsible Party: Principal Investigator, Yolradee Winuntamalakul, Principal Investigator, Navamindradhiraj University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 193/65 FB
Record Dates: First submitted 2023-12-01; First posted 2023-12-11 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Dry Age-related Macular Degeneration
MeSH Terms: interventions — Aspirin; Clopidogrel; Acetylcysteine

STUDY DESIGN:
Intervention Model Description: 1. Aspirin 81 mg/d or Clopidogrel 75 mg/d
  2. Aspirin 81 mg/d or Clopidogrel 75 mg/d with N-acetylcysteine 600 mg/d
  3. No medication
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Antiplatelet drug (Active Comparator): In this study, antiplatelet drugs are medications that patients take to treat their underlying condition, such as aspirin 81 mg/day or clopidogrel 75 mg/day.
  Interventions: Drug: Aspirin 81Mg Ec Tab; Drug: Clopidogrel
- Antiplatelet drug with antioxidant (Experimental): Antiplatelet drugs are medications that patients take to treat their underlying condition, such as aspirin 81 mg/day or clopidogrel 75 mg/day combined with N-acetylcysteine 600 mg/day.
  Interventions: Drug: Aspirin 81Mg Ec Tab; Drug: Clopidogrel; Drug: N-acetylcysteine
- No medication (No Intervention): Patient with no medication used.

INTERVENTIONS:
Drug: Aspirin 81Mg Ec Tab — Patients take aspirin 81 mg per day.
  Arms: Antiplatelet drug; Antiplatelet drug with antioxidant
Drug: Clopidogrel — Patients take clopidogrel 75 mg per day.
  Arms: Antiplatelet drug; Antiplatelet drug with antioxidant
Drug: N-acetylcysteine — Patients are given N-acetylcysteine 600 mg per day.
  Other Names: NAC-long
  Arms: Antiplatelet drug with antioxidant

SUMMARY:
The aim of this clinical trial is to evaluate the effect of low doses of antiplatelet medications (aspirin 81 mg/day or clopidogrel 75 mg/day) with or without a combination of antioxidants (N-acetylcysteine 600 mg/day) in a dry AMD patient with large drusen.

Participants will divided in to three groups.

* Participants who were already taking low dose antiplatelet medications.
* Participants who take the antiplatelet drug mentioned above in addition to the antioxidant prescribed by the investigator
* Participants does not use any medications.

ELIGIBILITY:
Inclusion Criteria:

* Dry AMD with at least 1 large drusen. According to the AREDS study, large drusen have a size of more than 125 micron.
* Patients can evaluate SD-OCT (Spectral domain optical coherence tomography), OCT angiography, and best-corrected visual acuity.
* Age range: 50-85 years
* Patients who have previously used antiplatelet drugs.

Exclusion Criteria:

* Patient with advanced AMD, such as geographic atrophy, neovascular complications (choroidal neovascularization)
* Patient with additional retinal diseases that affect visual acuity, e.g., retinal detachment, diabetic macular edema.
* Patient with a history of intravitreal anti-VEGF injection or macular laser.
* Patient using SSRIs, SNRIs, azole, NSAIDs, dual antiplatelet, anticoagulant medications.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Drusen volume analysis | 1 year
  To assess AMD progression in patient with large drusen, drusen volume was measured and analyzed in each patient group by OCT scan

SECONDARY OUTCOMES:
Best-corrected visual acuity change | 1 year
  To evaluate Best-corrected visual acuity in each patient group by ETDRS chart
Rate of disease progression | 1 year
  To evaluate disease progression to geographic atrophy or neovascular AMD by OCT scan and fundus photo
Side effects of medications intake | 1 year
  To evaluate the safety of the medication used by questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Department of ophthalmology, Faculty of medicine, Vajira hospital, Navamindradhiraj University, Bangkok, Dusit, Thailand

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-03-15): https://cdn.clinicaltrials.gov/large-docs/68/NCT06165068/Prot_SAP_ICF_000.pdf